CLINICAL TRIAL: NCT02804620
Title: From Clinic to Community: Using Peer Support as a Transition Model for Improving Long-term Diabetes-related Health Outcomes
Brief Title: From Clinic to Community Study
Acronym: C2C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Tricia Tang, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H14-02419
Record Dates: First submitted 2016-01-06; First posted 2016-06-17 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Peer Support; Diabetes Self-management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLEASED (Experimental): The PLEASED intervention arm will receive peer leader who is patients with diabetes that has been gone through our trainings. Also, they will receive three free health screenings (baseline, 3 months, 12 months) and monetary compensation for their time and effort.
  Interventions: Behavioral: Peer-led, Empowerment-based Approach to Self-management efforts in Diabetes
- Wait List (No Intervention): The wait list will receive three free health screening (at baseline, 3months, 12 months) and monetary compensation for their time and effort.

INTERVENTIONS:
Behavioral: Peer-led, Empowerment-based Approach to Self-management efforts in Diabetes — The investigators will train patients with type 2 diabetes who are well-controlled and pair them up with participants. Peer leaders will help the participants overcome their problems and teach them how to make changes by 5 step goal setting strategy. The peer leaders never give advice on any medical condition. All the medical questions will be referred to the research team.
  Other Names: PLEASED
  Arms: PLEASED

SUMMARY:
This study is a 12-month study. There are two different groups in the study. Both groups will enter the study after the graduation from 8-hour diabetes education course taught at VGH, St. Paul's, or Richmond Hospital. The first group will receive on-going support from their peers who have diabetes and are trained specifically to help other patients with diabetes. The second group will receive the usual care.

DETAILED DESCRIPTION:
This two-phase study is a randomized controlled trial (RCT) comparing usual care to a 12-month peer-led DSMS intervention designed to improve long-term diabetes-related health outcomes.

In Phase 1, the research team will implement a 30-hour peer leader training (PLT) program recruiting adults with type 2 diabetes and equipping them with the diabetes knowledge, facilitation strategies, and communication skills to deliver a DSMS intervention. In Phase 2, the researchers will conduct the peer support intervention, referred to as the Peer-Led, Empowerment-based Approach to Self-management Efforts in Diabetes (PLEASED). Patients randomized to the PLEASED arm will be paired with a peer leader and receive 12 weekly contacts (face-to-face and telephone support) from their peer leader (PL) in the first 3 months followed by 18 bi-weekly telephone support contacts over the last 9 months.

The goal of the PLEASED intervention is to help patients improve glycemic control and diabetes specific QOL and sustain these health benefits over the long-term. To achieve this goal, PLs will address 3 key functions of peer support that include assisting patients in the daily management of their diabetes, providing social and emotional support, and linking patients to clinical care resources.

Participants' inclusion criteria are: to (1) have type 2 diabetes, (2) be 21 years, (3) speak English or Vietnamese or any languages that their peer leaders speak, (4) be willing to be matched with a peer leader, and (5) have a personal land line telephone or mobile phone.

Peer leaders' inclusion criteria are: (1) have diabetes, (2) be 21 years, (3) speak English, (4) have transportation to attend training, (5) be willing to commit to a 30-hour training program, and (6) have a land line telephone or mobile phone (7) have a self-reported HbA1c of 8% or less.

ELIGIBILITY:
Inclusion Criteria for Participants:

* To be eligible for the study, patients have to:

  1. have type 2 diabetes,
  2. be 21 years,
  3. speak English or Vietnamese or any languages that their peer leaders speak,
  4. be willing to be matched with a peer leader, and
  5. have a personal land line telephone or mobile phone.

Exclusion Criteria for Participants:

* They should not participate in the study if they have physical limitations, serious health conditions or addictions to alcohol or drugs, which would hinder meaningful participation in the study.

Inclusion Criteria for Peer Leaders:

1. have diabetes,
2. be 21 years,
3. speak English,
4. have transportation to attend training,
5. be willing to commit to a 30-hour training program, and
6. have a land line telephone or mobile phone
7. have a self-reported HbA1c of 8% or less..

Exclusion Criteria for Peer Leaders:

* They should not participate in the study if they have physical limitations, serious health conditions or addictions to alcohol or drugs, which would hinder meaningful participation in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2014-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c% | 0, 3, 12 month(s)

SECONDARY OUTCOMES:
ApoB | 0, 3, 12 month(s)

OTHER OUTCOMES:
Change in diabetes-specific QoL | 0, 3, 12 month(s)
Blood Pressure | 0, 3, 12 month(s)
Height | 0, 3, 12 month(s)
Weight | 0, 3, 12 month(s)

CONTACTS AND LOCATIONS:
Overall Officials: Tricia S Tang, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norris SL, Nichols PJ, Caspersen CJ, Glasgow RE, Engelgau MM, Jack L, Snyder SR, Carande-Kulis VG, Isham G, Garfield S, Briss P, McCulloch D. Increasing diabetes self-management education in community settings. A systematic review. Am J Prev Med. 2002 May;22(4 Suppl):39-66. doi: 10.1016/s0749-3797(02)00424-5. PMID 11985934
- [Background] Padgett D, Mumford E, Hynes M, Carter R. Meta-analysis of the effects of educational and psychosocial interventions on management of diabetes mellitus. J Clin Epidemiol. 1988;41(10):1007-30. doi: 10.1016/0895-4356(88)90040-6. PMID 3193136
- [Background] Deakin T, McShane CE, Cade JE, Williams RD. Group based training for self-management strategies in people with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003417. doi: 10.1002/14651858.CD003417.pub2. PMID 15846663
- [Background] Effect of intensive diabetes treatment on the development and progression of long-term complications in adolescents with insulin-dependent diabetes mellitus: Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. J Pediatr. 1994 Aug;125(2):177-88. doi: 10.1016/s0022-3476(94)70190-3. PMID 8040759
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Haas L, Maryniuk M, Beck J, Cox CE, Duker P, Edwards L, Fisher EB, Hanson L, Kent D, Kolb L, McLaughlin S, Orzeck E, Piette JD, Rhinehart AS, Rothman R, Sklaroff S, Tomky D, Youssef G; 2012 Standards Revision Task Force. National standards for diabetes self-management education and support. Diabetes Care. 2013 Jan;36 Suppl 1(Suppl 1):S100-8. doi: 10.2337/dc13-S100. No abstract available. PMID 23264420
- [Background] Anderson G, Horvath J. The growing burden of chronic disease in America. Public Health Rep. 2004 May-Jun;119(3):263-70. doi: 10.1016/j.phr.2004.04.005. No abstract available. PMID 15158105
- [Background] Fischman J. Who will take care of you? US News World Rep. 2005 Jan 31-Feb 7;138(4):44-6. No abstract available. PMID 15700601
- [Background] Institute of Medicine of the National Academies (report). Crossing the quality chasm: A new heart system for the 21st century/Committee on Quality Health Care in America. Washington, DC. National Academy Press, 2001.
- [Background] Institute of Medicine (US) Committee on Understanding and Eliminating Racial and Ethnic Disparities in Health Care; Smedley BD, Stith AY, Nelson AR, editors. Unequal Treatment: Confronting Racial and Ethnic Disparities in Health Care. Washington (DC): National Academies Press (US); 2003. Available from http://www.ncbi.nlm.nih.gov/books/NBK220358/ PMID 25032386
- [Background] Reported by Joanne Currie, Executive Director of Canadian Diabetes Educators Certification Board.
- [Background] Lewin S, Munabi-Babigumira S, Glenton C, Daniels K, Bosch-Capblanch X, van Wyk BE, Odgaard-Jensen J, Johansen M, Aja GN, Zwarenstein M, Scheel IB. Lay health workers in primary and community health care for maternal and child health and the management of infectious diseases. Cochrane Database Syst Rev. 2010 Mar 17;2010(3):CD004015. doi: 10.1002/14651858.CD004015.pub3. PMID 20238326
- [Background] Dennis CL. Peer support within a health care context: a concept analysis. Int J Nurs Stud. 2003 Mar;40(3):321-32. doi: 10.1016/s0020-7489(02)00092-5. PMID 12605954
- [Background] Report of a World Health Organization consultation. Peer support programmes in diabetes November 5-7, 2007.
- [Background] Dale JR, Williams SM, Bowyer V. What is the effect of peer support on diabetes outcomes in adults? A systematic review. Diabet Med. 2012 Nov;29(11):1361-77. doi: 10.1111/j.1464-5491.2012.03749.x. PMID 22804713
- [Background] Smith SM, Paul G, Kelly A, Whitford DL, O'Shea E, O'Dowd T. Peer support for patients with type 2 diabetes: cluster randomised controlled trial. BMJ. 2011 Feb 15;342:d715. doi: 10.1136/bmj.d715. PMID 21324992
- [Background] Lorig K, Ritter PL, Laurent DD, Plant K, Green M, Jernigan VB, Case S. Online diabetes self-management program: a randomized study. Diabetes Care. 2010 Jun;33(6):1275-81. doi: 10.2337/dc09-2153. Epub 2010 Mar 18. PMID 20299481
- [Background] Dale J, Caramlau I, Sturt J, Friede T, Walker R. Telephone peer-delivered intervention for diabetes motivation and support: the telecare exploratory RCT. Patient Educ Couns. 2009 Apr;75(1):91-8. doi: 10.1016/j.pec.2008.09.014. Epub 2008 Nov 14. PMID 19013741
- [Background] Cade JE, Kirk SF, Nelson P, Hollins L, Deakin T, Greenwood DC, Harvey EL. Can peer educators influence healthy eating in people with diabetes? Results of a randomized controlled trial. Diabet Med. 2009 Oct;26(10):1048-54. doi: 10.1111/j.1464-5491.2009.02808.x. PMID 19900238
- [Background] Lorig K, Ritter PL, Villa FJ, Armas J. Community-based peer-led diabetes self-management: a randomized trial. Diabetes Educ. 2009 Jul-Aug;35(4):641-51. doi: 10.1177/0145721709335006. Epub 2009 Apr 30. PMID 19407333
- [Background] Murrock CJ, Higgins PA, Killion C. Dance and peer support to improve diabetes outcomes in African American women. Diabetes Educ. 2009 Nov-Dec;35(6):995-1003. doi: 10.1177/0145721709343322. Epub 2009 Sep 23. PMID 19776334
- [Background] Lorig K, Ritter PL, Villa F, Piette JD. Spanish diabetes self-management with and without automated telephone reinforcement: two randomized trials. Diabetes Care. 2008 Mar;31(3):408-14. doi: 10.2337/dc07-1313. Epub 2007 Dec 20. PMID 18096810
- [Background] Anderson-Loftin W, Barnett S, Bunn P, Sullivan P, Hussey J, Tavakoli A. Soul food light: culturally competent diabetes education. Diabetes Educ. 2005 Jul-Aug;31(4):555-63. doi: 10.1177/0145721705278948. PMID 16100331
- [Background] Keyserling TC, Samuel-Hodge CD, Ammerman AS, Ainsworth BE, Henriquez-Roldan CF, Elasy TA, Skelly AH, Johnston LF, Bangdiwala SI. A randomized trial of an intervention to improve self-care behaviors of African-American women with type 2 diabetes: impact on physical activity. Diabetes Care. 2002 Sep;25(9):1576-83. doi: 10.2337/diacare.25.9.1576. PMID 12196430
- [Background] Pratt C, Wilson W, Leklem J, Kingsley L. Peer support and nutrition education for older adults with diabetes. J Nutr Elder. 1987 Summer;6(4):31-43. doi: 10.1300/J052v06n04_04. No abstract available. PMID 3656067
- [Background] Heisler M, Vijan S, Makki F, Piette JD. Diabetes control with reciprocal peer support versus nurse care management: a randomized trial. Ann Intern Med. 2010 Oct 19;153(8):507-15. doi: 10.7326/0003-4819-153-8-201010190-00007. PMID 20956707
- [Background] Baksi AK, Al-Mrayat M, Hogan D, Whittingstall E, Wilson P, Wex J. Peer advisers compared with specialist health professionals in delivering a training programme on self-management to people with diabetes: a randomized controlled trial. Diabet Med. 2008 Sep;25(9):1076-82. doi: 10.1111/j.1464-5491.2008.02542.x. PMID 18937675
- [Background] McKay HG, Glasgow RE, Feil EG, Boles SM, Barrera M. Internet-based diabetes self-management and support: Initial outcomes from the Diabetes Network project, Rehabil Psychol 2002;47:31-48.
- [Background] Glasgow RE, Boles SM, McKay HG, Feil EG, Barrera M Jr. The D-Net diabetes self-management program: long-term implementation, outcomes, and generalization results. Prev Med. 2003 Apr;36(4):410-9. doi: 10.1016/s0091-7435(02)00056-7. PMID 12649049
- [Background] Thom DH, Ghorob A, Hessler D, De Vore D, Chen E, Bodenheimer TA. Impact of peer health coaching on glycemic control in low-income patients with diabetes: a randomized controlled trial. Ann Fam Med. 2013 Mar-Apr;11(2):137-44. doi: 10.1370/afm.1443. PMID 23508600
- [Background] Siminerio L, Ruppert KM, Gabbay RA. Who can provide diabetes self-management support in primary care? Findings from a randomized controlled trial. Diabetes Educ. 2013 Sep-Oct;39(5):705-13. doi: 10.1177/0145721713492570. Epub 2013 Jun 19. PMID 23782622
- [Background] Philis-Tsimikas A, Fortmann A, Lleva-Ocana L, Walker C, Gallo LC. Peer-led diabetes education programs in high-risk Mexican Americans improve glycemic control compared with standard approaches: a Project Dulce promotora randomized trial. Diabetes Care. 2011 Sep;34(9):1926-31. doi: 10.2337/dc10-2081. Epub 2011 Jul 20. PMID 21775748
- [Background] Gillespie P, O'Shea E, Paul G, O'Dowd T, Smith SM. Cost effectiveness of peer support for type 2 diabetes. Int J Technol Assess Health Care. 2012 Jan;28(1):3-11. doi: 10.1017/S0266462311000663. PMID 22617733
- [Background] Tang TS, Funnell M, Sinco B, Piatt G, Palmisano G, Spencer MS, Kieffer EC, Heisler M. Comparative effectiveness of peer leaders and community health workers in diabetes self-management support: results of a randomized controlled trial. Diabetes Care. 2014 Jun;37(6):1525-34. doi: 10.2337/dc13-2161. Epub 2014 Apr 10. PMID 24722495
- [Background] Tang TS, Funnell MM, Gillard M, Nwankwo R, Heisler M. The development of a pilot training program for peer leaders in diabetes: process and content. Diabetes Educ. 2011 Jan-Feb;37(1):67-77. doi: 10.1177/0145721710387308. Epub 2011 Jan 10. PMID 21220362
- [Background] Tang TS, Funnell MM, Gillard M, Nwankwo R, Heisler M. Training peers to provide ongoing diabetes self-management support (DSMS): results from a pilot study. Patient Educ Couns. 2011 Nov;85(2):160-8. doi: 10.1016/j.pec.2010.12.013. Epub 2011 Feb 2. PMID 21292425
- [Background] Tang TS, Sohal PS, Garg AK. Evaluating a diabetes self-management support peer leader training programme for the English- and Punjabi-speaking South-Asian community in Vancouver. Diabet Med. 2013 Jun;30(6):746-52. doi: 10.1111/dme.12179. Epub 2013 Apr 17. PMID 23506520
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Esliger DW, Tremblay MS. Technical reliability assessment of three accelerometer models in a mechanical setup. Med Sci Sports Exerc. 2006 Dec;38(12):2173-81. doi: 10.1249/01.mss.0000239394.55461.08. PMID 17146326
- [Background] Block G, Gillespie C, Rosenbaum EH, Jenson C. A rapid food screener to assess fat and fruit and vegetable intake. Am J Prev Med. 2000 May;18(4):284-8. doi: 10.1016/s0749-3797(00)00119-7. PMID 10788730
- [Background] Sarason I, Sarason B, Brock D, Pierce G. Social support: current status, current issues. Spielberger CE. Stress and Emotion: Anxiety, Anger, and Curiously. Washington DC: Taylor and Francis; 1998
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Resnicow K, Campbell M, Carr C, McCarty F, Wang T, Periasamy S, Rahotep S, Doyle C, Williams A, Stables G. Body and soul. A dietary intervention conducted through African-American churches. Am J Prev Med. 2004 Aug;27(2):97-105. doi: 10.1016/j.amepre.2004.04.009. PMID 15261895
- [Background] Abbey A, Abramis D, Caplan R. Effects of different sources of social support and social conflict on emotional well-being. Soc Sci Med 1985;6:2:111-129.
- [Background] Kulzer B, Hermanns N, Reinecker H, Haak T. Effects of self-management training in Type 2 diabetes: a randomized, prospective trial. Diabet Med. 2007 Apr;24(4):415-23. doi: 10.1111/j.1464-5491.2007.02089.x. Epub 2007 Feb 12. PMID 17298590
- [Result] Canadian Diabetes Association. The prevalence and costs of diabetes. Diabetes.ca (accessed December 1, 2013).
- [Result] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Result] Norris SL, Engelgau MM, Narayan KM. Effectiveness of self-management training in type 2 diabetes: a systematic review of randomized controlled trials. Diabetes Care. 2001 Mar;24(3):561-87. doi: 10.2337/diacare.24.3.561. PMID 11289485
- [Derived] Seddigh S, Tang TS. Social support and diabetes distress: Does the messenger matter as much as the message? Chronic Illn. 2023 Sep;19(3):681-685. doi: 10.1177/17423953221102622. Epub 2022 May 26. PMID 35619542
- [Derived] Afshar R, Askari AS, Sidhu R, Cox S, Sherifali D, Camp PG, Tang TS. Out of the mouths of Peer Leaders: Perspectives on how to improve a telephone-based peer support intervention in type 2 diabetes. Diabet Med. 2022 Sep;39(9):e14853. doi: 10.1111/dme.14853. Epub 2022 Apr 30. PMID 35437815